CLINICAL TRIAL: NCT00361114
Title: Efficacy of Sulphadoxine/Pyrimethamine and Chlorproguanil/Dapsone in 6-59 Month Old Children With Uncomplicated Malaria and in 2-10 Month Old Asymptomatic Infants.
Brief Title: IPT and Efficacy of Sulphadoxine/Pyrimethamine and Chlorproguanil/Dapsone in 6-59 Month Old Children With Malaria.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: SP arms were stopped due to high levels of treatment failure.CD not available.
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIF 35
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; chloroguanil, dapsone drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): SP in symptomatic children aged 6-59 months
  Interventions: Drug: sulphadoxine/pyrimethamine
- B (Experimental): SP to asymptomatic infected children aged 2-10 months
  Interventions: Drug: Sulfadoxine/pyrimethamine
- C (Experimental): Chlorproguanil/dapsone in symptomatic 6-59 month old children
  Interventions: Drug: Chlorproguanil/dapsone

INTERVENTIONS:
Drug: sulphadoxine/pyrimethamine — Sulfadoxine/pyremethamine (SP) given as a single dose per manufacturers recommendation (tablets 500mg sulphadoxine and 15mg pyremethamine; child's body weight 5-10Kgs ½ tablet, 11-20Kgs 1 tablet, 21-30 Kgs 1 ½ tablets)
  Other Names: Fansidar
  Arms: A
Drug: Chlorproguanil/dapsone — Chlorproguanil/ dapsone (CD) given daily for 3 days per manufacturers recommendations (tablets chlorproguanil 15mg/ dapsone 18.75 mg; 5-7.9Kgs 1 tablet, 8-11.9 Kg 1 ½ tablets, 12-15.9 2 tablets, 16-20.9 Kgs 2 ½ tablets, 21- 40Kg 5 tablets).
  Other Names: Lapdap
  Arms: C
Drug: Sulfadoxine/pyrimethamine — Sulfadoxine/pyremethamine (SP) given as a single dose per manufacturers recommendation (tablets 500mg sulphadoxine and 15mg pyremethamine; child's body weight 5-10Kgs ½ tablet, 11-20Kgs 1 tablet, 21-30 Kgs 1 ½ tablets)
  Other Names: Fansidar
  Arms: B

SUMMARY:
Intermittent Preventive Treatment of malaria in infants is a promising strategy to reduce incidence of clinical malaria in children under the age of 1 year. It is likely to be implemented as a malaria control strategy in Tanzania using sulfadoxine/pyremethamine SP. SP is failing as a first line treatment for clinical episodes of malaria and government policy is driving a change to use Artemesin Combination Therapy (ACT). The main ongoing Kilimanjaro IPTi study is looking at alternatives to SP for use in IPTi. Currently, as there is no evidence for the use of other drugs for IPT, SP will be continued for IPT in pregnancy and in infants. This study proposes to measure the efficacy of SP and chlorproguanil/dapsone (CD), in symptomatic 6- 59 month old children using standard methodology. These are both study drugs in the main IPTi study. This will help us to see how the efficacies of SP and CD in sick children relate to the efficacies for treating asymptomatic children with IPTi. In addition this proposal aims to test the efficacy of SP given to 2-10 month old asymptomatic infants (the target group for IPTi). Evidence suggests that asymptomatic malaria infections with low parasitaemia have a higher cure rate than symptomatic infections with high parasitaemia even when markers of resistance are highly prevalent. This second study aims to quantify this difference and will produce evidence to help policy makers know when drugs used for IPTi should be changed. Both studies will be open label and run concurrently in Hale, Korogwe district near to the main Kilimanjaro IPTi site in Tanzania.

DETAILED DESCRIPTION:
Introduction and Rational

This is part of a multicentre trial looking into antimalarial resistance within a series of Intermittent Preventive Treatment of malaria in Infants (IPTi) studies. IPTi is a promising intervention to reduce malaria in infants in malaria endemic countries. 3 doses of antimalarial drugs are given in the first year of life to asymptomatic infants at the time of 2nd and 3rd Diptheria, Tetanus and Pertusus immunisation and again at 9 months of age at time of measles immunisation. In the current Kilimanjaro IPTi study we are comparing 3 antimalarials (Mefloquine MQ, sulfadoxine/pyremethamine SP and chlorproguanil/dapsone CD) against placebo for IPTi in 2 transmission zones. Two published studies using SP for IPTi have shown different efficacies for this intervention. The first study (Schellenberg et al 2001) showed a 62% reduction in clinical cases of malaria and the second (Chandramohan et al, 2005) showed only a 25% reduction in clinical cases of malaria. The two sites differ in several ways, the first was carried out in an area of moderate to low transmission with a moderate rate of SP resistance in Tanzania and the latter was carried out in an area of intense but seasonal malaria with a low rate of SP resistance in Ghana. The current IPTi study is being carried out in a site of high transmission with expected high rates of SP resistance. Data from a site 100km away indicates SP efficacy to be 55% (Mutabingwa et al, 2001). There is no data on SP or other study drugs at the ongoing study sites.

In addition there is evidence (Personal communication Chandramohan 2005) that the outcome (Adequate Parasite Response (APR)) of asymptomatic parasitaemia in infants is better than that in symptomatic 6-59 month old children when using SP. For this reason we plan a novel study examining the efficacy of SP in asymptomatic 2-10 month old infants, the target age group for IPTi.

The main objective of this component of the drug resistance study is to understand the relationship between the efficacy of antimalarial drugs used for IPTi and the long term effect of IPTi on incidence of clinical malaria. Schellenberg et al (2005). observed a 36% reduction in the incidence of clinical malaria in the second year of life in the SP IPTi group compared to the placebo group even though the last course of SP IPTi was given at 9 months of age (Schellenberg et al, 2005). This suggests that SP IPTi in an area with moderate malaria transmission and moderate levels of resistance to SP (+/-25%) IPTi may enhance the development of immunity against malaria. In contrast, a study in Ghana in area with very high and seasonal malaria transmission and very low resistance to SP (<10%) showed a 20% increase in the incidence of clinical malaria with high parasite density (>5000 parasites/ml) in SP IPTi group compared to placebo group. The nature of the relationship between drug resistance and the long term effect of IPTi on malaria remains unclear.

Parasite clearance rate depends on the efficacy of antimalarial drug and host immunity. Host immunity depends on age - immunity in infants is likely to be lower than the immunity in 1-4 year old children. Parasite clearance rate depends on parasite density, multiplicity of infection, and the type of host response - these factors differ between clinical episodes of malaria and asymptomatic parasitaemia. The interaction between antimalarial drug and host response during a clinical episode of malaria is likely to be different from that during asymptomatic malaria parasitaemia. Although infants with mild illness will not be excluded from IPTi administration at routine EPI clinics, the majority of infants will be asymptomatic when they receive IPTi. Thus results of the standard WHO in vivo drug sensitivity studies conducted in 6-59 month-old symptomatic children are unlikely to be applicable to 2-10 month old mostly asymptomatic infants receiving IPTi. However, there is no empirical evidence to support or refute this assertion.

In order to understand the relationship between level of drug resistance and long terms effects of IPTi, the exact level of drug resistance in the IPTi target infants needs to be established and related to IPTi efficacy. Thus a modified WHO in vivo drug resistance study in 2-10 month old asymptomatic infants needs to be conducted as part of the Kilimanjaro IPTi study and a comparison made with the efficacy of SP estimated from a standard WHO 6-59 month WHO in vivo efficacy study.

Objectives

We therefore propose 2 studies that have the following objectives:

1. Enumerate the drug efficacies of SP and CD in the study area using the standard WHO in vivo drug efficacy methodology in symptomatic children aged 6-59 months,
2. Enumerate the efficacy of SP in asymptomatic 2-10 month olds using a modified WHO in vivo drug efficacy methodology, the target population for IPTi and
3. Determine the difference of efficacy when using SP for the different indications, ie between its use in symptomatic and asymptomatic children.

Methods

Study 1 is a standard in vivo WHO drug efficacy study looking at parasite positive symptomatic children between the ages of 6 and 59 months treated with SP or CD. They will be followed up after 1,2 3, 7,14,21 and 28 days. At each visit a blood slide and filter paper will be collected. Endpoints are day 28 recrudescence rates.

Study 2 is a modified in vivo drug efficacy study in the age group directly affected by IPTi, namely 2-10 months of age. Asymptomatic children will be followed up at days 1, 2, 3,7,14, 21 and 28 only. Endpoint is day 28 recrudescence rate. Blood slide and filter paper will only be taken on day 7, 14 and 28 unless the child has a fever or has reported fever in the last 48 hours.

Sample size and study subjects

Table 1 Study Arm Expected (assumed) rate of adequate parasitological response by day 28 (APR) Acceptable 95% confidence limit (precision) Sample Size needed based on expected APR and acceptable precision Total sample size (corrected for assumed 10% loss to follow-up and 10% nonadherence) 6-59 month symptomatic children SP 60% +/-6% 292* 330 CD 805 +/-7.5% 131 145

2-10 month asymptomatic children SP 75% +/-7.5% 146* 161

*SP study numbers are calculated to detect a 15% difference of APR by day 28 between symptomatic 6-59 month old children and asymptomatic 2-10 month old children with 80% power at the 5% significance level using a ratio of 2 symptomatic cases to 1 asymptomatic case.

Children attending a single health dispensary (Hale dispensary, Korogwe District,Tanga Region, Tanzania) aged between 6-59 months with a fever or history of fever within the preceding 48 hours will be asked to take part. If they fit the entry criteria (see attached protocol) and consent, they will be enrolled in the standard WHO in vivo efficacy study. Asymptomatic children aged between 2 and 10 months attending the MCH clinic for immunisations and weighing will be invited to take part in the 2-10 month efficacy study and those eligible for the study and consenting will be enrolled into the study.

Study Site

The project will take place in Hale Dispensary, a government dispensary offering primary care and MCH services to a population of more than 8,000, with an average of 30 new births a month. Hale is situated in Korogwe district,Tanga region, northeastern Tanzania and is lowland with high malaria transmission. It is less than 10 km from the IPTi study site.

Ethical considerations

It is expected that first line antimalarial drug policy will change in November 2006 from SP to lumefantrine/arthemeter. After this date it will not be ethical to continue the 6-59 month study in symptomatic children. However for the asymptomatic children it will be ethical to continue as SP use continues in asymptomatic women for IPTp and if adopted as a strategy for Tanzania, SP will be used for IPTi. Therefore we plan to carry out the SP efficacy in 6-59 month study in symptomatic children as soon as possible and if the national policy changes before completion of the study we will have to halt it. The 2-10 month old asymptomatic study will run concurrently until completion.

In the study the second line drug will be lumefantrine/arthemeter for all children should treatment fail.

Clinical safety of subjects is paramount. We will encourage mothers to bring their children for review during the follow up period when ever the child is sick. We have budgeted for a transport allowance for the mothers to help them make the journey when necessary. We will ensure 24 hour access to a member of the study team at all time. This person will be able to call on medical staff covering all clinical trial activities in Korogwe District Hospital for advice and possible emergency transfer to the hospital and assessment. An emergency vehicle is on standby 24 hours a day.

ELIGIBILITY:
For 6-59 month study

Inclusion Criteria:

* Aged 6-59 months
* Weight of 4.5 Kgs or greater.
* Not enrolled in IPTi trial
* Absence of severe malnutrition (defined as a child whose weight-for-height is below 3 standard deviations of less than 70% of the median of WHO reference values, or who has symmetrical edema involving at least the feet)
* A slide-confirmed infection with P. falciparum only
* Initial parasite density between 2,000 and 200,000 asexual parasites per microliter.
* Absence of general danger signs among children < 5 years (see below) Measured axillary temperature ³37.5 °C
* Ability to attend stipulated follow-up visits
* Informed consent provided by parent/guardian
* Absence of history of hypersensitivity reactions to any of the drugs being evaluated

Exclusion Criteria:

* Enrolled in IPTi trial
* Severe malnutrition (defined as above)
* No slide confirmed infection with P. falciparum
* Initial parasite density < 2,000 or > 200,000 asexual parasites per microliter.
* Presence of general danger signs among children < 5 years (inability to drink or breastfeed; vomiting everything; recent history of convulsions; lethargy or unconsciousness; inability to sit or stand up) or other signs of severe and complicated falciparum malaria according to WHO definitions
* Measured axillary temperature <37.5 °C
* Inability to attend stipulated follow-up visits
* Informed consent not provided by parent/guardian
* History of hypersensitivity reactions to any of the drugs being evaluated

For 2-10 month study

Inclusion criteria.

* Aged 2-10 months
* Weight of 4.5 Kgs or greater.
* Not enrolled in IPTi trial
* Absence of severe malnutrition
* A slide-confirmed infection with P. falciparum only
* Any parasite density assessed by research microscopists.
* Absence of general danger signs among children < 5 years (inability to drink or breastfeed; vomiting everything; recent history of convulsions; lethargy or unconsciousness; inability to sit or stand up) or other signs of severe and complicated falciparum malaria according to WHO definitions
* Measured axillary temperature < 37.5 °C
* Ability to attend stipulated follow-up visits
* Informed consent provided by parent/guardian
* Absence of history of hypersensitivity reactions to SP.

Exclusion criteria are not listed separately in the WHO protocol, as they are the opposite of the inclusion criteria.

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2006-07; Primary Completion 2007-08 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Clinical /Parasitological Outcomes (WHO 2003) | Day 14 and 28
Early Treatment Failure (ETF) | 3 days
§ Development of danger signs or severe malaria on Day 1, 2, or 3, in the presence of parasitemia | 3 Days
§ Parasitemia on Day 2 higher than Day 0 count irrespective of axillary temperature | 2 nd day
§ Parasitemia on Day 3 with axillary temperature ≥37.5°C | 3 rd day
§ Parasitemia on Day 3 ≥ 25% of count on Day 0 | 3 rd Day
Late Clinical Failure (LCF) | After Day 3 to day 28
§ Development of danger signs or severe malaria from Day 4 to Day 28 in the presence of parasitemia, without previously meeting any of the criteria of ETF | Day 4 - 28
§ Presence of parasitemia and axillary temperature ≥37.5° C on any day from Day 4 to Day 28, without previously meeting any of the criteria of ETF | Day 4 to Day 28
Late parasitological failure (LPF) - | Day 4 - 28
Presence of parasitemia on Day 14, 21, or 28 and axillary temperature <37.5°C without previously meeting any of the criteria of ETF or LCF (after exclusion of re-infection by PCR for failures at days 14-28) | Day 14, 21, or 28
Adequate Clinical and Parasitological Response (ACPR) - | Day 28
Absence of parasitemia on Day 28 irrespective of axillary temperature, without previously meeting any of the criteria of ETF, LCF or LPF | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Roly D Gosling, MD, Principal Investigator — London School of Hygiene and Tropical Medicine; Samwel Gesase, MD, Principal Investigator — National Institute of Medical Research, Tanzania; Jaqueline Mosha, MD, Principal Investigator — Kilimanjaro Christian Medical College, Tanzania
Locations (1):
- Hale Dispensary, Korogwe, Tanga, Tanzania

REFERENCES:
- [Derived] Gesase S, Gosling RD, Hashim R, Ord R, Naidoo I, Madebe R, Mosha JF, Joho A, Mandia V, Mrema H, Mapunda E, Savael Z, Lemnge M, Mosha FW, Greenwood B, Roper C, Chandramohan D. High resistance of Plasmodium falciparum to sulphadoxine/pyrimethamine in northern Tanzania and the emergence of dhps resistance mutation at Codon 581. PLoS One. 2009;4(2):e4569. doi: 10.1371/journal.pone.0004569. Epub 2009 Feb 24. PMID 19238219